CLINICAL TRIAL: NCT03875781
Title: Non Inferiority Multicenter Phase III Randomized Trial Comparing Preoperative Chemotherapy Only to Chemotherapy Followed by Chemoradiotherapy for Locally Advanced Resectable Rectal Cancer (Intergroup FRENCH-GRECCAR- PRODIGE)
Brief Title: Non Inferiority Study of Preoperative Chemotherapy Without Pelvic Irradiation for Rectal Cancer
Acronym: NORAD01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P170920J
Record Dates: First submitted 2019-02-18; First posted 2019-03-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer; Advanced Cancer
Keywords: Rectal cancer; FOLFIRINOX,; chemotherapy; radiochemotherapy; surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: To demonstrate the non inferiority of preoperative modified FOLFIRINOX chemotherapy compared to radiochemotherapy in primary resectable locally advanced rectal cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Modified Folfirinox (Experimental): Experimental : preoperative chemotherapy:
  Modified FOLFIRINOX regimen comprised oxaliplatin 85mg/m2 + irinotecan 180mg/m2 + Folinic acid 400 mg/m2 at day1, then 5-FU given as a continuous infusion over 46h every two weeks. Six cycles are planned preoperatively.
  Interventions: Drug: Chemotherapy
- B: Modified Folfirinox followed by Radiochemotherapy (Active Comparator): Active comparator: preoperative chemotherapy : Modified FOLFIRINOX regimen comprised oxaliplatin 85mg/m2 + irinotecan 180mg/m2 + Folinic acid 400 mg/m2 at day1, then 5-FU given as a continuous infusion over 46h every two weeks. Six cycles are planned preoperatively FOLLOWED BY Preoperative radiochemotherapy with concurrent capecitabine 825 mg/m2/12h 5 days/week and intensity modulated radiation therapy using a simultaneous integrated boost technique with 45 Gy in 25 fractions in pelvic volume and 50 Gy in 25 fractions to the tumor
  Interventions: Drug: Radiochemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Arm A : Experimental
  * Intervention Type : Drug
  * Intervention Name : Modified FOLFIRINOX (experimental arm)
  * Intervention Description : preoperative chemotherapy: Modified FOLFIRINOX regimen comprised oxaliplatin 85mg/m2 + irinotecan 180mg/m2 + Folinic acid 400 mg/m2 at day1, then 5-FU given as a continuous infusion over 46h every two weeks. Six cycles are planned preoperatively.
  Arms: A: Modified Folfirinox
Drug: Radiochemotherapy — Arm B: Active comparator
  * Intervention Name : modified FOLFIRINOX followed by preoperative standardized radiochemotherapy (control arm)
  * Intervention Description : preoperative chemotherapy: Modified FOLFIRINOX regimen comprised oxaliplatin 85mg/m2 + irinotecan 180mg/m2 + Folinic acid 400 mg/m2 at day1, then 5-FU given as a continuous infusion over 46h every two weeks. Six cycles are planned preoperatively.followed by preoperative radiochemotherapy with concurrent capecitabine 825 mg/m2/12h 5 days/week and intensity modulated radiation therapy using a simultaneous integrated boost technique with 45 Gy in 25 fractions in pelvic volume and 50 Gy in 25 fractions to the tumor.
  Arms: B: Modified Folfirinox followed by Radiochemotherapy

SUMMARY:
This study is a non-inferiority phase III randomised trial comparing preoperative chemotherapy alone (modified FOLFIRINOX) to chemotherapy followed by chemoradiotherapy in patients with primary resectable locally advanced rectal cancer. The primary endpoint of the study is 3-year progression free survival.

Expected 3 year PFS rate in the preoperative chemotherapy followed by chemoradiotherapy arm is 75%. This hazard rate, in an exponential survival model, corresponds to a decrease in the 3-year PFS rate on the preoperative chemotherapy arm to 67%. The study will randomize 540 patients (270 in the chemotherapy group and 270 in the chemoradiotherapy group) in 42 french academic centers.

DETAILED DESCRIPTION:
This study is a national, multicenter, open-label randomized, 2-arm phase III non-inferiority trial.

Patients with mid or low LARC (cT3N0 or cT1-T3N+ with CRM > 2 mm on pretreatment MRI) will be randomized to two arms of treatment: one experimental arm with systemic FOLFIRINOX chemotherapy for 3 months and one control arm with systemic FOLFIRINOX chemotherapy for 3 months followed by conventional standardized radiochemotherapy (intensified-modulated radiotherapy 50Gy + capecitabine). The choice of FOLFIRINOX for preoperative chemotherapy is based on recent data regarding its safety and efficacy rectal cancer with or without metastatic disease. Since the annual world meeting of ASCO 2020, a new standard of treatment has been adopted using the combination of chemotherapy followed by radiochemotherapy that has been show to improve disease free survival in phase III controlled randomized trial (Conroy et al, J Clin Oncol 38: 2020 (suppl; abstr 4007).

All patients will have reassessment MRI after preoperative treatment and before surgery.

Objectives and study endpoints

- primary endpoint : 3-year progression-free survival (PFS) from the time to randomization. In this trial, a modified definition of PFS will be used for the primary endpoint. The rationale for using this modified definition of PFS is to better assess time to failure of the whole treatment strategy (preoperative treatment and surgery).

Progression will be assessed as follows:

* progression during preoperative treatment and before surgery: circumferential resection margin ≤ 2mm at MRI reeassessemnt and diagnosis of any new distant lesion whatever the site (liver, lung, peritoneum, adrenal) are considered as progression events.
* progression after surgery: recurrence/progression after surgery or death, whatever comes first.

  * Secondary endpoints: treatment related toxicity, treatment compliance, R0 resection rate, sphincter saving surgery rate, postoperative morbidity and mortality rates, loco-regional recurrence free survival, overall survival, bowel and sexual functions at diagnosis, quality of life, radiologic and pathologic response after preoperative treatment.

Statistical analysis A sample size of 518 patients, based on an expected accrual duration of 36 months, 60 months follow-up, and an expected 3 year PFS rate in the preoperative chemotherapy followed by chemoradiotherapy arm of 75%, is expected to provide 239 PFS events required to provide 80% power to declare non-inferiority of the preoperative chemotherapy arm when the true hazard ratio between arms is 1.0 (H1). This design has a global type one-error rate of 0.05 if the true hazard ratio between arms is 1.39 (H0). This hazard rate, in an exponential survival model, corresponds to a decrease in the 3-year PFS rate on the preoperative chemotherapy arm to 67%. By considering a rate of 4% for not informative or lost to follow-up patients the total number of patients to be included in this trial was 518*100/96 = 540 patients.

Ancillary studies Pronostic value of circulating cancer cells before and after preoperative treatment and after surgery in patients undergoing surgery for rectal cancer after chemotherapy or radiochemotherapy will be evaluated. After assessment of prognostic value of each rate on survival, recurrence and response to treatment, evaluation of prognostic impact of variation of the rate during differents phases of treatment will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven middle or low rectal carcinoma, ≤ 10 cm from the anal verge on MRI (sagittal slide)
* cT3N0 and/or cT1-T3N+ on pretreatment imaging work up (pelvic contrast enhanced MRI and/or endorectal ultrasound),
* Pretreatment predictive circumferential margin > 2mm on pretreatment imaging work up (pelvic contrast enhanced MRI)
* Patients must be 18 years old or older
* A World Health Organization (WHO/ECOG) performance status of 0 or 1
* Informed consent signed
* Patients of childbearing / reproductive potential should use adequate birth control measures during the study treatment period and for at least 6 months after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.

Exclusion Criteria:

* Rectal tumor > 10 cm from the anal verge on MRI (sagittal slide)
* cT4 tumor on pretreatment imaging work up (pelvic contrast enhanced MRI and/or endorectal ultrasound) or involvement of external sphincter
* Circumferential margin ≤ 2 mm on pretreatment imaging work up (pelvic contrast enhanced MRI)
* Metastatic disease
* Prior pelvic irradiation or any contraindication to pelvic irradiation
* Contraindication to oxaliplatin or irinotecan or 5FU based chemotherapy
* Concomitant treatment with warfarin is contraindicated and warafarin must be replaced whenever possible to allow for inclusion.
* Recent or concomitant treatment with brivudine is contraindicated
* contraindications to 5-FU: complete and permanent insufficiency in dihydropyrimidine dehydrogenase, bone marrow insufficiency, chronic and severe infection
* contraindication to irinotecan : inflammatory bowel disease, bilirubin serum level > 3 times the upper limit of the normal rate, severe bone marrow insufficiency, WHO/ECOG performence status > 2,
* Concomitant treatment with millepertuis.
* contraindication to oxaliplatin :

  *bone marrow insufficiency before treatment initiation (neutrophil count <2x109/L and/or platelet count <100x109/L), peripheral neuropathy with permanent invalidity before treatment initiation
* severe renal insufficiency (Creatinin clearance <30 ml/min)
* contraindications to folinic acid : Biermer anemia and other anemia related to B12 vitamin insufficiency
* contraindications to capecitabin : severe renal insufficiency (Creatinin clearance <30 ml/min), complete and permanent insufficiency in dihydropyrimidine dehydrogenase
* live attenuated vaccine should not be used during and 6 months after preoperative treatment.
* Previous colorectal cancer
* Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years
* Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* protected adults
* Pregnancy or breastfeeding
* Patient with no national health or universal plan affiliation coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2019-06-05 (Actual); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Survival | 3 years
  3-year progression-free survival

SECONDARY OUTCOMES:
Acute treatment toxicity | Up to 1 month after the end of preoperative treatment
  Acute and late treatment related toxicity: the rates of treatment related toxicity grade II or more
Late toxicity related to treatment | 3 years after surgery
  Late treatment related toxicity: the rates of treatment related toxicity grade II or more
Compliance to treatment | Up to 1 month after the end of preoperative treatment
  The rate of patients that receive full dose treatment
Radiological response | 28±5 days after the end of preoperative treatment
  Radiologic response on post-treatment MRI based on tumor size reduction and tumor regression grade (ymrTRG)
The rate of R0 resection | 4 weeks after surgery
  Rate of complete resection with safe > 1mm circumferential and longitudinal margin
Quality of mesorectal excision: 3-grades Quirke scoring system | 4 weeks after surgery
  3-grades Quirke scoring system of the quality of mesorectal excision
Number of lymph nodes harvested | 4 weeks after surgery
  A count of number of lymph nodes harvested
Size of circumferential margin | 4 weeks after surgery
  Mesurement of circumferential margin
Size of longitudinal margin | 4 weeks after surgery
  Mesurement of longitudinal margin
Sphincter saving surgery rate | 4 weeks after surgery
  The rate of surgery with intestinal continuity and anal sphincter preservation
Postoperative morbidity | 30 days after resection
  Postoperative morbidity: 30 day or in-hospital postoperative morbidity rates
Postoperative mortality | 30 days after resection
  Postoperative mortality: 30 day or in-hospital postoperative mortality rates
Pathologic response after chemotherapy | 4 weeks after surgery
  Pathologic response on Rodel Tumor Regression Grade
Pathologic response after chemoradiotherapy | 4 weeks after surgery
  Pathologic response after chemoradiotherapy: rate of major pathologic response base on Rodel Tumor Regression Grade
Loco-regional recurrence free survival | At 3 years
  Loco-regional recurrence free survival: 3-year locoregional recurrence free survival rates
Uncontrolled local recurrence | At 3 years
  Uncontrolled local recurrence: 3-year uncontrolled local recurrence free survival rates
Overall survival | At 3 years
  Overall survival: 3 year overall survival rates
Overall survival | At 5 years
  Overall survival: 5 year overall survival rates
EORTC QLQ-CR29 | Diagnosis time
  Assessed by the validated scales of quality of life for Colorectal Cancer Patients (QLQ-CR29) of the European Organisation for Research and Treatment of Cancer (EORTC). The scales ranges from 25 to 104 (104 is the worst quality of life)
EORTC QLQ-CR29 | 28±5 days after the end of preoperative treatment
  Assessed by the validated scales of quality of life for Colorectal Cancer Patients (QLQ-CR29) of the European Organisation for Research and Treatment of Cancer (EORTC). The scales ranges from 25 to 104 (104 is the worst quality of life)
EORTC QLQ-CR29 | At 6 months after surgery
  Assessed by the validated scales of quality of life for Colorectal Cancer Patients (QLQ-CR29) of the European Organisation for Research and Treatment of Cancer (EORTC). The scales ranges from 25 to 104 (104 is the worst quality of life)
EORTC QLQ-CR29 | 1 year after surgery
  Assessed by the validated scales of quality of life for Colorectal Cancer Patients (QLQ-CR29) of the European Organisation for Research and Treatment of Cancer (EORTC). The scales ranges from 25 to 104 (104 is the worst quality of life)
LARS Scores | Diagnosis time
  Bowel function assessed by the Low Anterior Resection Syndrome (LARS) score. The score ranges from 0 to 42 (42 is the most severe LARS)
LARS Scores | 28±5 days after the end of preoperative treatment
  Bowel function assessed by the Low Anterior Resection Syndrome (LARS) score. The score ranges from 0 to 42 (42 is the most severe LARS)
LARS Scores | 6 months after surgery
  Bowel function assessed by the Low Anterior Resection Syndrome (LARS) score. The score ranges from 0 to 42 (42 is the most severe LARS)
LARS Scores | 1 year after surgery
  Bowel function assessed by the Low Anterior Resection Syndrome (LARS) score. The score ranges from 0 to 42 (42 is the most severe LARS)
Quality of life - physical functioning: QLQ-C30 | At diagnosis
  Health related physical functioning assessed by the validated scale for Cancer Patients (QLQ-C30) of the European Organisation for Research and Treatment of Cancer (EORTC). The scales ranges from 0 to 100 (100 is the worst physical functioning)
Quality of life - physical functioning: QLQ-C30 | 28±5 days after the end of preoperative treatment
  Health related physical functioning assessed by the validated scale for Cancer Patients (QLQ-C30) of the European Organisation for Research and Treatment of Cancer (EORTC). The scales ranges from 0 to 100 (100 is the worst physical functioning)
Quality of life - physical functioning: QLQ-C30 | 6 months after surgery
  Health related physical functioning assessed by the validated scale for Cancer Patients (QLQ-C30) of the European Organisation for Research and Treatment of Cancer (EORTC). The scales ranges from 0 to 100 (100 is the worst physical functioning)
Quality of life - physical functioning: QLQ-C30 | 1 year after surgery
  Health related physical functioning assessed by the validated scale for Cancer Patients (QLQ-C30) of the European Organisation for Research and Treatment of Cancer (EORTC). The scales ranges from 0 to 100 (100 is the worst physical functioning)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane BENOIST, MD,PHD, Study Chair — Service de chirurgie digestive et oncologique Hôpital Bicêtre - 94275 LE KREMLIN BICETRE
Locations (1):
- BENOIST, Le Kremlin-Bicêtre, Île-de-France Region, France

REFERENCES:
- [Background] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Background] Wiltink LM, Chen TY, Nout RA, Kranenbarg EM, Fiocco M, Laurberg S, van de Velde CJ, Marijnen CA. Health-related quality of life 14 years after preoperative short-term radiotherapy and total mesorectal excision for rectal cancer: report of a multicenter randomised trial. Eur J Cancer. 2014 Sep;50(14):2390-8. doi: 10.1016/j.ejca.2014.06.020. Epub 2014 Jul 21. PMID 25060825
- [Background] Schrag D, Weiser MR, Goodman KA, Gonen M, Hollywood E, Cercek A, Reidy-Lagunes DL, Gollub MJ, Shia J, Guillem JG, Temple LK, Paty PB, Saltz LB. Neoadjuvant chemotherapy without routine use of radiation therapy for patients with locally advanced rectal cancer: a pilot trial. J Clin Oncol. 2014 Feb 20;32(6):513-8. doi: 10.1200/JCO.2013.51.7904. Epub 2014 Jan 13. PMID 24419115
- [Background] Bensignor T, Brouquet A, Dariane C, Thirot-Bidault A, Lazure T, Julie C, Nordlinger B, Penna C, Benoist S. Pathological response of locally advanced rectal cancer to preoperative chemotherapy without pelvic irradiation. Colorectal Dis. 2015 Jun;17(6):491-8. doi: 10.1111/codi.12879. PMID 25524450
- [Background] Deng Y, Chi P, Lan P, Wang L, Chen W, Cui L, Chen D, Cao J, Wei H, Peng X, Huang Z, Cai G, Zhao R, Huang Z, Xu L, Zhou H, Wei Y, Zhang H, Zheng J, Huang Y, Zhou Z, Cai Y, Kang L, Huang M, Peng J, Ren D, Wang J. Modified FOLFOX6 With or Without Radiation Versus Fluorouracil and Leucovorin With Radiation in Neoadjuvant Treatment of Locally Advanced Rectal Cancer: Initial Results of the Chinese FOWARC Multicenter, Open-Label, Randomized Three-Arm Phase III Trial. J Clin Oncol. 2016 Sep 20;34(27):3300-7. doi: 10.1200/JCO.2016.66.6198. Epub 2016 Aug 1. PMID 27480145
- [Derived] Brouquet A, Bachet JB, Huguet F, Karoui M, Artru P, Sabbagh C, Lefevre JH, Vernerey D, Mariette C, Vicaut E, Benoist S; on behalf the FRENCH , GRECCAR, PRODIGE study groups. NORAD01-GRECCAR16 multicenter phase III non-inferiority randomized trial comparing preoperative modified FOLFIRINOX without irradiation to radiochemotherapy for resectable locally advanced rectal cancer (intergroup FRENCH-GRECCAR- PRODIGE trial). BMC Cancer. 2020 May 29;20(1):485. doi: 10.1186/s12885-020-06968-1. PMID 32471382